CLINICAL TRIAL: NCT03381430
Title: A Open-label, One-arm Trial of Gefitinib Combined With Radiotherapy as Adjuvant Therapy in Completely Resected Patients With Pathological Stage IIIA-N2 Non-small Cell Lung Cancer Harbouring Sensitive Mutations of EGFR
Brief Title: Gefitinib Combine Radiotherapy as Therapy for Patients With NSCLC Harbouring Sensitive Mutations of EGFR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Collaborators: China-Japan Friendship Hospital (Other); Peking University Cancer Hospital & Institute (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRAY
Record Dates: First submitted 2017-11-15; First posted 2017-12-22 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gefitinib + Radiotherapy (Experimental): Experimental: Gefitinib Gefitinib 250 mg/day oral daily Radiotherapy Total dose 50-54Gy, divided dose 1.8-2Gy
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — Gefitinib 250 mg/day oral daily

SUMMARY:
To explore the survival benefit of the gefitinib combined with radiotherapy as adjuvant therapy for completely resected patients with Pathological stage IIIA-N2 NSCLC harbouring sensitive mutations of EGFR.

DETAILED DESCRIPTION:
Cisplatin-based adjuvant chemotherapy is standard of care for patients with stage II-IIIA non-small cell lung cancer (NSCLC). Activating somatic mutations of the tyrosine kinase domain of epidermal growth factor receptor (EGFR) have been characterized in a subset of patients with advanced NSCLC. The recently study of gefitinib (G) versus vinorelbine+cisplatin (VP) as adjuvant treatment in stage II-IIIA (N1-N2) NSCLC with EGFR-activating mutation (ADJUVANT)shows that G had significantly longer median DFS (28.7 months) than VP (18.0months). 3-year DFS was significantly better with G (34.0% vs 27.0%; p= 0.013) and subgroup analysis of patients treated with G, lymph node status (pN1/N2) demonstrated significant correlation with DFS.

At present, postoperative radiotherapy has been widely used in the treatment of all kinds of cancer, and the guidelines also recommend postoperative radiotherapy for stage IIIA-pN2 NSCLC. The retrospective study of Lee et. al. reported on the use of postoperative radiotherapy (PORT) as first strategy after resection of stage IIIA-pN2 NSCLC. The result showed that the five-year overall OS was significantly higher in patients treated with PORT and postoperative chemotherapy (POCT) than in patients treated with PORT alone. This open-label phase II trial is studying gefitinib combined with radiotherapy to see how well it works in treating patients who have undergone surgery for Pathological stage IIIA-N2 NSCLC with EGFR activating mutation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided.
* Males or females aged ≥18 years, < 75 years.
* Target population is completely resected pathological stage IIIA-N2 NSCLC with EGFR exon 19 deletions and exon 21 L858R activating mutation.
* Underwent radical resection
* The patient did not receive any neoadjuvant chemotherapy or EGFR-TKI targeted therapy before surgery
* Patient who can start the investigational therapy within 3-6 weeks after the complete resection
* ECOG performance status 0-1.
* Life expectancy ≥12 weeks.
* Adequate hematological function: Absolute neutrophil count (ANC) ≥2.0 x 109/L, and Platelet count ≥100 x 109/L, and Hemoglobin ≥9 g/dL (may be transfused to maintain or exceed this level).
* Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN), Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 x ULN in subjects without liver metastases; ≤ 5 x ULN in subjects with liver metastases.
* Adequate renal function: Serum creatinine ≤ 1.25 x ULN, or ≥ 60 ml/min.
* Female subjects should not be pregnant or breast-feeding.

Exclusion Criteria:

* Patients with prior exposure to agents directed at the HER axis (e.g. erlotinib, gefitinib, cetuximab, trastuzumab).
* Patients with prior any systemic chemotherapy, immunotherapy or biotherapy
* Known severe hypersensitivity to gefitinib or any of the excipients of this product.
* Patients with prior radiotherapy.
* Not fully recovered from the previous surgery.
* History of another malignancy in the last 5 years with the exception of the following: basal cell carcinoma of the skin and in situ carcinoma of the uterine cervix.
* Patients who harbouring exon 20 T790M mutation.
* Patient who has any active infection (e.g. acute pneumonia, hepatitis B or hepatitis C).
* Dysphagia or known malabsorption of drugs.
* Patient with serious heart, liver, kidney or other important organ dysfunction.
* Pregnancy or lactation women or women may be positive for pregnancy before the first medication.
* Patient has fertility but not willing to take contraceptive measures or whose sexual partners are unwilling to take contraceptive measures.
* Researcher believes the patient's condition is not suitable for the clinical study.
* Researcher judged the patient's lack of compliance with the study.
* Known severe hypersensitivity to gefitinib or any of the excipients of this product.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | CT scan, abdominal ultrasound every 3 months, brain MRI every 6 months, bone scan every 12 months for up to 3 years.
  From start of anti-cancer therapy until progression or death. To evaluate the disease free survival of gefitinib combined with radiotherapy as adjuvant therapy in completely resected patients with Pathological stage IIIA-pN2 NSCLC harbouring sensitive mutations of EGFR.Disease free survival (DFS)- defined as the time from initial medication to the first documented disease progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival | 6 years
  evaluated in the 6 years since treatment begain
3 yeas DFS rate | 3 years
  To compare the adjuvant treatment arm in terms of 3 yeas DFS rate.
5 years DFS rate | 5 years
  To compare the adjuvant treatment arm in terms of 5 years DFS rate.
5 years OS rate | 5 years
  To compare the adjuvant treatment arm in terms of 5 years OS rate.
Number of Participants with Adverse Events | In the period of Gefitinib 250 mg/day oral daily for 24 months. Radiotherapy total dose 50-54Gy, divided dose 1.8-2Gy.
  The safety and tolerability profile of gefitinib at a 250 mg daily dose relative to that of radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Guang-ying Zhu, MD, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, China